CLINICAL TRIAL: NCT04486625
Title: AN OPEN-LABEL, PARALLEL-GROUP, PHARMACOKINETIC STUDY OF MULTIPLE INTRAVENOUS DOSES OF AZTREONAM AND AVIBACTAM IN SUBJECTS WITH SEVERE RENAL IMPAIRMENT AND NORMAL RENAL FUNCTION
Brief Title: Pharmacokinetic Study of Aztreonam-Avibactam in Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C3601006
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2022-09

CONDITIONS: Renal Insufficiency
Keywords: Infection
MeSH Terms: conditions — Renal Insufficiency; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Normal renal function
  Interventions: Drug: Aztreonam-Avibactam
- Cohort 2 (Experimental): Severe renal impairment (not on dialysis)
  Interventions: Drug: Aztreonam-Avibactam

INTERVENTIONS:
Drug: Aztreonam-Avibactam — 500/167 mg ATM/AVI loading infusion, followed by 1500/500 mg ATM/AVI extended loading infusion, then 1500/500 mg ATM/AVI maintenance dose infusion every 6 hours
  Arms: Cohort 1
Drug: Aztreonam-Avibactam — 675/225 mg ATM/AVI loading infusion, followed by 675/225 mg ATM/AVI extended loading infusion, then 675/225 mg ATM/AVI maintenance dose infusion every 8 hours
  Arms: Cohort 2

SUMMARY:
This Phase 1 study is being conducted to evaluate the effect of severe renal impairment on the PK, safety and tolerability of Aztreonam-Avibactam. Results from this study along with previous renal impairment data from each of the Aztreonam-Avibactam components will be used to confirm the proposed dosing adjustment in severe renal impairment which was based on modelling/simulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects and/or male subjects between the ages of 18 and 75 years, inclusive. Male and female subjects of childbearing potential must agree to use highly effective method(s) of contraception
* Body mass index (BMI) of 17.5 to 40.5 kg/m2; and a total body weight >50 kg (110 lb)
* Stable renal function defined as </=25% difference between 2 measurements of eGFR obtained on 2 separate occasions during the screening period that are at least 72 hours but no more than 14 days apart Specific Requirements for Healthy Subjects with Normal Renal Function
* Normal renal function (eGFR>/= 80 mL/min) at Screening based on the Day -2 value, using the MDRD formula adjusting for BSA
* Demographically comparable to the group of subjects with severe impaired renal function Specific Requirements for Subjects with Severe Renal Impairment
* Good general health commensurate with the population with chronic kidney disease.
* Documented severe renal impairment indicated by eGFR >15 -</=30 mL/min but not requiring hemodialysis, using the MDRD formula adjusting for BSA

Exclusion Criteria:

* Positive urine drug test
* History of regular alcohol use (within 6 months) exceeding 7 drinks/week for female or 14 drinks/week for male subjects
* Treatment with an investigational product within 30 days or 5 half-lives preceding the first dose of investigational product (whichever is longer)
* Subjects with abnormalities in clinical laboratory tests (AST, ALT, Total bilirubin, aPTT, PT, INR) at Screening
* Pregnant females; breastfeeding females; fertile male subjects and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product. For subjects with severe renal impairment, concomitant medications may be given if considered necessary for the subject welfare (eg, standard therapy for underlying diseases), are not contraindicated with the study drug, and are unlikely to interfere with the PK/PD response of the study drug. Use of oral anticoagulants and potent inhibitors of OAT1 and/or OAT3 (eg, probenecid) are prohibited in all subjects.
* Blood donation (excluding plasma donations) of approximately 1 pint or more within 60 days prior to dosing
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* History of serious allergy, hypersensitivity or any serious reaction to aztreonam, carbapenem, monobactam or other beta-lactam antibiotics, avibactam, or any of the excipients of the respective (investigational) medicinal products
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Other acute or chronic medical or psychiatric condition
* Past or current history of epilepsy or seizure disorders excluding febrile seizures of childhood Exclusion criteria: Subjects with Severe Renal Impairment
* Any significant hepatic, cardiac, or pulmonary disease
* Renal allograft recipients or subjects who are clinically nephrotic
* Subjects requiring dialysis
* Screening supine 12-lead ECG demonstrating QT interval corrected by Fridericia's formula (QTcF) >470 msec or a QRS interval >120 msec
* Screening supine BP >/=180 millimeters of mercury (mm Hg) (systolic) or >/=110 mm Hg (diastolic), on a single measurement (confirmed by a single repeat, if necessary) following at least 5 minutes of rest Exclusion criteria: Subjects with Normal Renal Function
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including clinically relevant and significant drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Screening supine 12-lead ECG demonstrating QTcF >450 msec or a QRS interval >120 msec
* Screening supine BP >/=140 mm Hg (systolic) or >/=90 mm Hg (diastolic), following at least 5 minutes of supine rest

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3601006

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a Phase 1, open-label, parallel-group study where an intravenous (IV) loading dose (30-minute infusion) followed by multiple IV doses (3-hour infusion) of aztreonam-avibactam (ATM-AVI) were administered to participants with severe renal impairment (not on dialysis) (Cohort 1) and to healthy participants with normal renal function (Cohort 2).
Groups:
- Cohort 1: Normal Renal Function: Participants with normal renal function received 30-minute IV loading dose infusion (500/167 mg aztreonam [ATM]/avibactam [AVI]), followed by 3-hour IV extended loading infusion (1500/500 mg ATM/AVI), then 3-hour 1500/500 mg ATM/AVI maintenance dose infusion every 6 hours on Days 1 to 3.
- Cohort 2: Severe Renal Impairment: Participants with severe renal impairment (not on dialysis) received 30-minute IV loading dose infusion (675/255 mg aztreonam [ATM]/avibactam [AVI]), followed by 3-hour IV extended loading infusion (675/255 mg ATM/AVI), then 3-hour 675/255 mg ATM/AVI maintenance dose infusion every 8 hours on Days 1 to 3.
Period: Overall Study
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean | 61.0 (1.67) | 67.8 (8.56) | 64.1 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 4 | 5 | 9
  Race: Black or African American | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 0
  Ethnicity: Not Hispanic or Latino | 6 | 5 | 11
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 98.65 (6.354) | 101.06 (13.068) | 99.75 (9.491)

OUTCOME MEASURES:

1. Primary Outcome: Total Daily Area Under the Plasma Concentration-time Profile From Time 0 to 24 Hours at Steady-state (AUC0-24,ss) of Aztreonam (ATM)
Description: AUC0-24,ss of ATM in Cohort 1 was calculated by 4*AUC0-tau (tau = 6 hours), where AUC0-tau was area under the concentration-time profile from time 0 to time tau (the dosing interval). AUC0-24,ss of ATM in Cohort 2 was calculated by 3*AUC0-tau (tau = 8 hours), where AUC0-tau was area under the plasma concentration-time profile from time 0 to time tau (the dosing interval).
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: The analysis population included all participants treated with study medication who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*hour per milliliter (ug*hr/mL)
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Microgram*hour per milliliter (ug*hr/mL) | 922.9 (16) | 733.5 (16)
Statistical Analysis 1: Comparison: Cohort 1: Normal Renal Function vs Cohort 2: Severe Renal Impairment; Test type: Other — Analysis of variance (ANOVA) was used to compare the natural log transformed AUC0-24,ss between the normal renal function group (Reference) and the severe renal impairment group (Test). The geometric least squares mean point estimate and the associated 90% confidence intervals (CIs) for the difference of each comparison was estimated; Ratio (%) of adjusted geometric means = 79.48, 90% CI 2-sided [66.52 to 94.96]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of ATM
Description: The Cmax of ATM was observed directly from data.
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (ug/mL)
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Microgram per milliliter (ug/mL) | 57.34 (13) | 43.34 (11)
Statistical Analysis 1: Comparison: Cohort 1: Normal Renal Function vs Cohort 2: Severe Renal Impairment; Test type: Other — ANOVA was used to compare the natural log transformed Cmax between the normal renal function group (Reference) and the severe renal impairment group (Test). The geometric least squares mean point estimate and the associated 90% CIs for the difference of each comparison was estimated; Ratio (%) of adjusted geometric means = 75.58, 90% CI 2-sided [66.10 to 86.43]

3. Primary Outcome: AUC0-24,ss of Avibactam (AVI)
Description: AUC0-24,ss of AVI in Cohort 1 was calculated by 4*AUC0-tau (tau = 6 hours), where AUC0-tau was area under the concentration-time profile from time 0 to time tau (the dosing interval). AUC0-24,ss of AVI in Cohort 2 was calculated by 3*AUC0-tau (tau = 8 hours), where AUC0-tau was area under the plasma concentration-time profile from time 0 to time tau (the dosing interval).
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
ug*hr/mL | 164.8 (18) | 204.6 (20)
Statistical Analysis 1: Comparison: Cohort 1: Normal Renal Function vs Cohort 2: Severe Renal Impairment; Test type: Other — ANOVA was used to compare the natural log transformed AUC0-24,ss between the normal renal function group (Reference) and the severe renal impairment group (Test). The geometric least squares mean point estimate and the associated 90% CIs for the difference of each comparison was estimated; Ratio (%) of of adjusted geometric means = 124.19, 90% CI 2-sided [100.18 to 153.97]

4. Primary Outcome: Cmax of AVI
Description: The Cmax of AVI was observed directly from data.
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
ug/mL | 11.08 (14) | 11.35 (14)
Statistical Analysis 1: Comparison: Cohort 1: Normal Renal Function vs Cohort 2: Severe Renal Impairment; Test type: Other — [test comment as in outcome 2, analysis 1]; Ratio (%) of adjusted geometric means = 102.42, 90% CI 2-sided [87.55 to 119.83]

5. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to Time Tau (The Dosing Interval)(AUC0-tau) of ATM
Description: The AUC0-tau was calculated by linear/log trapezoidal method. The dosing interval (tau) was 6 hours for normal renal function (Cohort 1) and 8 hours for severe renal impairment (Cohort 2).
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
ug*hr/mL | 230.8 (16) | 244.3 (16)

6. Secondary Outcome: Time for Cmax (Tmax) of ATM
Description: The Tmax was observed directly from data as time of first occurrence.
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Hours | 2.92 [2 to 2.92] | 2.92 [2.92 to 3.75]

7. Secondary Outcome: Observed Plasma Concentration at the End of the Dosing Interval (Tau) (Ctau) of ATM
Description: The Ctau was observed directly from data. The dosing interval (tau) was 6 hours for normal renal function (Cohort 1) and 8 hours for severe renal impairment (Cohort 2).
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
ug/mL | 21.43 (19) | 18.55 (24)

8. Secondary Outcome: Terminal Elimination Half-life (t1/2) of ATM
Description: The t1/2 was calculated by loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log linear concentration time curve. Only those data points judged to describe the terminal log linear decline were used in the regression.
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Hours | 2.605 (0.34944) | 4.902 (1.4286)

9. Secondary Outcome: Clearance (CL) of ATM
Description: The CL was calculated by dose/AUC0-tau, where AUC0-tau was area under the concentration-time profile from time 0 to time tau (the dosing interval). The dosing interval (tau) was 6 hours for normal renal function (Cohort 1) and 8 hours for severe renal impairment (Cohort 2).
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/hr)
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Liters per hour (L/hr) | 6.499 (16) | 2.761 (16)

10. Secondary Outcome: Renal Clearance (CLr) of ATM
Description: The CLr was calculated by Ae0-tau/AUC0-tau, where Ae0-tau was cumulative amount of drug recovered unchanged in urine up to time tau and AUC0-tau was area under the plasma concentration time profile from time 0 to time tau (the dosing interval). The dosing interval (tau) was 6 hours for normal renal function (Cohort 1) and 8 hours for severe renal impairment (Cohort 2).
Time Frame: In Cohort 1, at predose on Day 3, during 0-2, 2-4, and 4-6 hours after the start of a maintenance dose infusion. In Cohort 2, at predose on Day 3, during 0-2, 2-4, 4-6, and 6-8 hours after the start of a maintenance dose infusion.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
L/hr | 4.527 (18) | 1.477 (23)

11. Secondary Outcome: Apparent Volume of Distribution (Vz) of ATM
Description: The Vz was calculated by dose/(AUC0-tau*kel), where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve and AUC0-tau was area under the concentration-time profile from time 0 to time tau (the dosing interval). The dosing interval (tau) was 6 hours for the normal renal function group (Cohort 1) and 8 hours for the severe renal impairment group (Cohort 2).
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Liters (L) | 24.25 (23) | 18.79 (21)

12. Secondary Outcome: Apparent Volume of Distribution at Steady-state (Vss) of ATM
Description: Vss was calculated by CL*MRT, where CL was clearance and MRT was mean residence time.
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
L | 23.70 (29) | 18.46 (19)

13. Secondary Outcome: Cumulative Amount of Drug Recovered Unchanged in Urine up to Time Tau (Ae0-tau) of ATM
Description: The Ae0-tau was the sum of (urine concentration*sample volume). The dosing interval (tau) was 6 hours for normal renal function (Cohort 1) and 8 hours for severe renal impairment (Cohort 2).
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram (mg)
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Milligram (mg) | 1047 (11) | 361.2 (19)

14. Secondary Outcome: Percent of Dose Recovered Unchanged in Urine up to Time Tau (Ae0-tau%) of ATM
Description: The Ae0-tau was calculated by 100*Ae0-tau/dose, where Ae0-tau was cumulative amount of drug recovered unchanged in urine up to time tau. The dosing interval (tau) was 6 hours for normal renal function (Cohort 1) and 8 hours for severe renal impairment (Cohort 2).
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent of dose
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Percent of dose | 69.68 (11) | 53.51 (19)

15. Secondary Outcome: AUC0-tau of AVI
Description: The UC0-tau was calculated by linear/log trapezoidal method. The dosing interval (tau) was 6 hours for normal renal function (Cohort 1) and 8 hours for severe renal impairment (Cohort 2).A
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
ug*hr/mL | 41.19 (18) | 68.31 (20)

16. Secondary Outcome: Tmax of AVI
Description: The Tmax was observed directly from data as time of first occurrence.
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Hours | 2.46 [2 to 2.92] | 2.92 [2 to 3.25]

17. Secondary Outcome: Ctau of AVI
Description: as for outcome 7
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
ug/mL | 3.100 (24) | 5.597 (39)

18. Secondary Outcome: t1/2 of AVI
Description: as for outcome 8
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Hours | 3.188 (0.071391) | 6.524 (1.6469)

19. Secondary Outcome: CL of AVI
Description: The CL was calculated by dose/AUC0-tau, where AUC0-tau was area under the plasma concentration-time profile from time 0 to to time tau (the dosing interval). The dosing interval (tau) was 6 hours for normal renal function (Cohort 1) and 8 hours for severe renal impairment (Cohort 2).
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
L/hr | 12.16 (18) | 3.295 (20)

20. Secondary Outcome: CLr of AVI
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
L/hr | 11.30 (20) | 3.948 (36)

21. Secondary Outcome: Vz of AVI
Description: as for outcome 11
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
L | 55.83 (19) | 30.14 (16)

22. Secondary Outcome: Vss of AVI
Description: Vss was calculated by CL*MRT, where CL was clearance and MRT was mean residence time.
Time Frame: Predose, 2, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 16, and 24 hours after start of a maintenance dose infusion on Day 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
L | 37.37 (30) | 27.78 (16)

23. Secondary Outcome: Ae0-tau of AVI
Description: as for outcome 13
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
mg | 465.6 (11) | 270.0 (17)

24. Secondary Outcome: Ae0-tau% of AVI
Description: as for outcome 14
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent of dose
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Percent of dose | 93.19 (11) | 119.9 (17)

25. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) (All-causality)
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a product; the event need not necessarily have a causal relationship with the treatment or usage. A serious adverse event is any untoward medical occurrence at any dose that: (1) results in death; (2) is life threatening (immediate risk of death); (3) requires inpatient hospitalization or prolongation of existing hospitalization; (4) results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); (5) results in congenital anomaly/birth defect; or that is considered to be an important medical event. Treatment-emergent are events between first dose of study medication and up to at least 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. A severe AE is defined as a event interferes significantly with participant's usual function.
Time Frame: Day 1 up to at least 28 days after last dose of study medication (maximum of 33 days).
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Participants
  Participants with AEs | 2 | 3
  Participants with serious AEs | 0 | 0
  Participants with severe AEs | 0 | 0
  Participants discontinued from study due to AEs | 0 | 0
  Participants discontinued study drug due to AEs and continue study | 0 | 0
  Participants with dose reduced or temporary discontinuation due to AEs | 0 | 0

26. Secondary Outcome: Number of Participants With TEAEs (Treatment-related)
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a product; the event attributed to the study medication. A serious AE is any untoward medical occurrence at any dose that: (1) results in death; (2) is life threatening (immediate risk of death); (3) requires inpatient hospitalization or prolongation of existing hospitalization; (4) results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); (5) results in congenital anomaly/birth defect; or that is considered to be an important medical event. Treatment-emergent are events between first dose of study medication and up to at least 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. A severe AE is defined as a event interferes significantly with participant's usual function.
Time Frame: Day 1 up to at least 28 days after last dose of study medication (maximum of 33 days).
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Participants
  Participants with AEs | 0 | 3
  Participants with serious AEs | 0 | 0
  Participants with severe AEs | 0 | 0
  Participants discontinued from study due to AEs | 0 | 0
  Participants discontinued study drug due to AEs and continue study | 0 | 0
  Participants with dose reduced or temporary discontinuation due to AEs | 0 | 0

27. Secondary Outcome: Number of Participants With Categorical Post-Baseline Vital Signs Data
Description: Categorical post-baseline vital signs included: (1) pulse rate: value less than (<) 40 beats per minute (bpm), lager than (>) 120 bpm; (2) supine diastolic blood pressure (DBP): value <50 mmHg, change of more than or equal to (>=) 20 mmHg increase, change of >=20 mmHg decrease; (3) supine systolic blood pressure (SBP): value <90 mmHg, change of >=30 mmHg increase, change of >=30 mmHg decrease.
Time Frame: Days 1 to 3
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Participants
  Pulse rate <40 bpm | 0 | 0
  Pulse rate >120 bpm | 0 | 0
  Supine DBP <50 mmHg | 0 | 0
  Supine DBP change >=20 mmHg increase | 0 | 0
  Supine DBP change >=20 mmHg decrease | 0 | 0
  Supine SBP <90 mmHg | 0 | 0
  Supine SBP change >=30 mmHg increase | 0 | 1
  Supine SBP change >=30 mmHg decrease | 0 | 0

28. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG)
Description: Criteria for ECG abnormalities: maximum QT interval >500 milliseconds (msec); maximum QTc interval of >=450 msec to less than or equal to (<=) 480 msec, >480 msec, and >500 msec and a maximum change of <30 change<=60 or >60 msec from baseline; maximum QTcF (Fridericia's Correction) interval of >=450 msec to <=480 msec, >480 msec, and >500 msec and a maximum change of <30 change<=60 or >60 msec from baseline.
Time Frame: Days 1 to 3
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Participants
  QT interval value > 500 msec | 0 | 0
  450 msec<= QTc interval value <=480 msec | 0 | 2
  QTc interval value >480 msec | 0 | 0
  QTc interval value >500 msec | 0 | 0
  30 msec< QTc interval change <=60 msec | 0 | 0
  QTc interval change >60 msec | 0 | 0
  450 msec<= QTcF interval value <=480 msec | 0 | 2
  QTcF interval value >480 msec | 0 | 0
  QTcF interval value >500 msec | 0 | 0
  30 msec< QTcF interval change <=60 msec | 0 | 0
  QTcF interval change >60 msec | 0 | 0

29. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Following laboratory parameters were abnormal (without regard to baseline abnormality): hemoglobin, hematocrit, erythrocytes, lymphocytes, neutrophils, activated partial thromboplastin time, protein, urea nitrogen, creatinine, urate, urine glucose, and urine protein.
Time Frame: Days 1 to 3
Population: The analysis population included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
Number analyzed (Participants) | 6 | 5
Participants
  Hemoglobin (gram per deciliter [g/dL]) <0.8*lower limit of normal (LLN) | 0 | 3
  Hematocrit (%) <0.8*LLN | 0 | 3
  Erythrocytes (10^6 per cubic millimeter [10^6/mm^3]) <0.8*LLN | 0 | 4
  Lymphocytes (10^3 per cubic millimeter [10^3/mm^3]) <0.8*LLN | 0 | 1
  Neutrophils (10^3/mm^3) >1.2*upper limit of normal (ULN) | 0 | 1
  Activated partial thromboplastin time (second) >1.1*ULN | 0 | 1
  Protein (g/dL) <0.8*LLN | 0 | 1
  Urea Nitrogen (milligram per deciliter [mg/dL]) >1.3*ULN | 0 | 5
  Creatinine (mg/dL) >1.3*ULN | 0 | 5
  Urate (mg/dL) >1.2*ULN | 0 | 3
  Urine glucose (mg/dL) >=1 | 0 | 3
  Urine protein (mg/dL) >=1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 up to at least 28 days after last dose of study drug (maximum of 33 days).
Description: Participants were only counted once per treatment for each category.
Arm/Group | Cohort 1: Normal Renal Function | Cohort 2: Severe Renal Impairment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 2/6 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Normal Renal Function (N=6) | Cohort 2: Severe Renal Impairment (N=5)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT04486625/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT04486625/SAP_001.pdf